CLINICAL TRIAL: NCT05250804
Title: The Effect of Helfer Skin Tap Technique on Pain, Fear, and Anxiety in Children Undergoing Intramuscular Injection: Randomized Controlled Trial
Brief Title: The Effect of Helfer Skin Tap Technique on Pain, Fear, and Anxiety in Children Undergoing Intramuscular Injection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aylin Kurt (Other)
Responsible Party: Sponsor-Investigator, Aylin Kurt, Principal Investigator, Bartın Unıversity
Organization: Bartın Unıversity (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: 2021-SBB-0513
Record Dates: First submitted 2022-01-28; First posted 2022-02-22 (Actual); Last update posted 2023-05-11 (Actual); Status verified 2023-05

CONDITIONS: Pain, Acute; Fear Anxiety; Child, Only; Injection Site
MeSH Terms: conditions — Acute Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): All registered participants in the intervention group, will receive the intramuscular injection with Helfer Skin Tap Technique.
  Interventions: Other: Helfer Skin Tap Technique
- No intervention (No Intervention): All registered participants in the intervention group, will receive the intramuscular injection with Routine Technique. Routine Technique involved inserting the injection intra muscularly at 90 degree angle into Dorso gluteal muscles without tapping after cleaning with alcohol swab.

INTERVENTIONS:
Other: Helfer Skin Tap Technique — Helfer Skin Tap Technique is a technique in which the researcher taps the Dorso gluteal muscle by counting 1-15 with the palmar aspect of fingers (non-dominant hand) in rhythmic manner before inserting the injection intra muscularly at 90 degree and remove the needle quickly again by tapping and counting 1-3.
  Arms: Experimental

SUMMARY:
The aim of this study was to examine the effect of the Helfer Skin Tapping technique on pain, fear, and anxiety in children who received intramuscular injections.

The research hypotheses are as follows:

H0: There is no significant difference between the intervention group and the the control group in the mean score of the "Wong-Baker FACES Pain Rating Scale", "Child Fear Scale", and "Child Anxiety Scale-State" during and after the Helfer Skin Tapping technique.

H1: During and after the Helfer Skin Tapping technique, the mean score of the "Wong-Baker FACES Pain Rating Scale", "Child Fear Scale", and "Child Anxiety Scale-State" is significantly lower in the intervention group compared to the control group.

DETAILED DESCRIPTION:
In this study, there will be two groups as the intervention (who will receive an intramuscular injection with the Helfer Skin Tapping technique) and the control group (who will receive an intramuscular injection with Routine Technique). A power analysis was performed based on the number of children in both groups, based on another study using the scales to be used in the research. According to the calculations made in the G-Power 3.1 Demo package program, when the effect size was accepted as 0.8, it was seen that at least 32 cases in each group would be sufficient for 80% power. Children who meet the research criteria will be randomly assigned to the intervention and control groups via http://www.randomize.org/ by assigning a number to the order of arrival at the hospital. The intramuscular injection will be applied to both the intervention and control groups. The children in the intervention group will receive an intramuscular injection with the Helfer Skin Tapping technique and the control group will receive an intramuscular injection with Routine Technique in the pediatric emergency service. A researcher and a nurse were employed for the intramuscular injection both for the intervention and control groups. A pediatric nurse performed the intramuscular injection for all children and the other researcher helped the children to assess their pain, fear, and anxiety level. Pain, fear, and anxiety in children were evaluated by the children and their parents before, during, 5 minute after the procedure. The intramuscular injection will be performed by the same nurse both in the intervention and control groups.

ELIGIBILITY:
Inclusion Criteria:

* The child is between the ages of 4-10
* The child's application to the Pediatric Emergency Unit
* Parent and child agreeing to participate in the project
* Absence of speech and visual impairment of the child and his parents

Exclusion Criteria:

* The child is not between the ages of 4-10
* The child's application to another department except for the Pediatric Emergency Unit
* Parent and child not agreeing to participate in the project
* Having speech and visual impairment of the child and his parents

Ages: 4 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 64 (Actual)
Dates: Start 2022-02-28 (Actual); Primary Completion 2022-07-12 (Actual); Study Completion 2022-07-12 (Actual)

PRIMARY OUTCOMES:
Difference of the mean score of the "Wong Baker FACES Pain Rating Scale" between intervention and control groups | 12 months
  "Wong Baker FACES Pain Rating Scale" will be completed intramuscular injection with Helfer Skin Tap Technique that gathers quantitative data that will pain about intramuscular injection in children. A minimum of 0 points and a maximum of 10 points can be obtained from the scale. The higher scores mean the higher pain. This scale will also be completed at during and 5. minutes after the intervention. The quantitative data will be used to measure a change in the children's pain level before, and after the proposed intervention. The scale will be made with Routine Technique in the control group. At the end of the study, the change of the mean score of "Wong-Baker FACES Pain Rating Scale" between intervention and control groups will be examined. Data will be analyzed using Statistical Package for the Social Sciences package program.
Difference between the mean score of the "Child Fear Scale" between intervention and control groups | 12 months
  "The Child Fear Scale" will be completed intramuscular injection with Helfer Skin Tap Technique that gathers quantitative data that will fear about the intramuscular injection in children. A minimum of 0 points and a maximum of 20 points can be obtained from the scale. The higher scores mean the higher fear. This scale will also be completed at during and 5 minutes after the intervention. The quantitative data will be used to measure a change in the children's fear level before, and after the proposed intervention. The scale will be made with Routine Technique in the control group. At the end of the study, the change of the mean score of "The Child Fear Scale" between intervention and control groups will be examined. Data will be analyzed using Statistical Package for the Social Sciences package program.
Difference between the mean score of the "Child Anxiety Meter-State" between intervention and control groups | 12 months
  "The Child Anxiety Meter-State" will be completed intramuscular injection with Helfer Skin Tap Technique that gathers quantitative data that will anxiety about the intramuscular injection in children. A minimum of 0 points and a maximum of 10 points can be obtained from the scale. The higher scores mean the higher anxiety. This scale will also be completed at during and 5 minutes after the intervention. The quantitative data will be used to measure a change in the children's anxiety level before and after the proposed intervention. The scale will be made with Routine Technique in the control group. At the end of the study, the change of the mean score of "The Child Anxiety Meter-State" between intervention and control groups will be examined. The Child Anxiety Meter-State total score mean of the children in the intervention group will be lower after the intervention compared to the control group. Data will be analyzed using Statistical Package for the Social Sciences package program.

SECONDARY OUTCOMES:
Change of the mean scores obtained by the children in the intervention group from the "Wong Baker FACES Pain Rating Scale" before and after the intervention. | 12 months
  "The Wong Baker FACES Pain Rating Scale" will be completed before intramuscular injection with Helfer Skin Tap Technique that gathers quantitative data that will address pain about the inhaler treatment with a nebulizer in children.A minimum of 0 points and a maximum of 10 points can be obtained from the scale. The higher scores mean the higher pain. This scale will also be completed at the intervention during and during and 5 minutes after the intervention. The quantitative data will be used to measure the change in the children's pain before, and after the proposed intervention. Data will be analyzed using Statistical Package for the Social Sciences package program.
Change of the mean scores obtained by the children in the intervention group from the "Child Fear Scale" before and after the intervention. | 12 months
  "The Child Fear Scale" will be completed before intramuscular injection with Helfer Skin Tap Technique that gathers quantitative data that will address fear about the inhaler treatment with a nebulizer in children. A minimum of 0 points and a maximum of 20 points can be obtained from the scale. The higher scores mean the higher fear. This scale will also be completed at the intervention during and 1. minutes after the intervention. The quantitative data will be used to measure the change in the children's fear before, and after the proposed intervention. Data will be analyzed using Statistical Package for the Social Sciences package program.
Change of the mean scores obtained by the children in the intervention group from the " Child Anxiety Meter-State " before and after the intervention. | 12 months
  "The Child Anxiety Meter-State" will be completed before intramuscular injection with Helfer Skin Tap Technique that gathers quantitative data that will address anxiety about the inhaler treatment with a nebulizer in children. A minimum of 0 points and a maximum of 10 points can be obtained from the scale. The higher scores mean the higher anxiety. This scale will also be completed at the intervention during and 1. minutes after the intervention. The quantitative data will be used to measure the change in the children's anxiety before, and after the proposed intervention. Data will be analyzed using Statistical Package for the Social Sciences package program.

CONTACTS AND LOCATIONS:
Locations (1):
- Bartın University, Bartın, Province, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol
Time Frame: 12 months